CLINICAL TRIAL: NCT07191821
Title: Modulation of Endothelial Function in Alzheimer's Disease by 18kDa Translocator Protein
Brief Title: TSPO Modulation in AD
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 23/LO/0080
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer s Disease
MeSH Terms: interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The first 6 participants will participate in an open label safety phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XBD173 followed by Placebo (Other): Participants will receive experimental medication XBD173 twice a day for 4 weeks followed by a 6 week washout before beginning a 4 week course of placebo twice a day. Both arms are double blinded
  Interventions: Drug: XBD173
- Placebo followed by XBD173 (Other): Participants will receive placebo twice a day for 4 weeks followed by a 6 week washout before beginning a 4 week course of experimental medication XBD173 twice a day. Both arms are double blinded
  Interventions: Drug: XBD173

INTERVENTIONS:
Drug: XBD173 — Small molecule experimental medication binding to mitochondrial protein TSPO

SUMMARY:
The aim of this study is to determine whether pharmacological modulation of TSPO (with XBD173, 90mg twice daily, orally, for 28 days) improves neurovascular coupling (NVC) in AD relative to placebo. The main questions it aims to answer are:

Does pharmacological modulation of TSPO (with XBD173, 90mg twice daily, orally, for 28 days) improve neurovascular coupling (NVC) in people with AD compared to placebo? NVC will be defined as the change in hippocampal cerebral blood flow (CBF) that follows a memory task (ΔCBF(h)).

Does pharmacological modulation of TSPO (with XBD173, 90mg twice daily, orally, for 28 days): Increase cerebral blood flow (CBF); Reduce blood brain barrier leak (rate and volume) determined by Gd enhanced DCE-MRI; Increase plasma Amyloid 40/42; Reduce soluble markers of endothelial cell activation(sVCAM1, sICAM1, PECAM1, E-selectin, vWF); Improve markers of peripheral endothelial cell function; Cerebrovascular reactivity in response to CO2 inhalation

The first six participants will undergo a dose escalation phase. The first 3 participants will receive XBD173 (90mg, once daily, 28 days) and the subsequent 3 participants will receive XBD173 (90mg, twice daily, 28 days). This phase will be open label. Participants will have 1 safety visits and 2 assessment visits. Each Assessment visit will involve clinical tests, a blood test and an MRI scan. Participants in the Randomisation phase participants will be given either 90mg of XBD173, twice daily or a placebo (dummy drug) for 4 weeks, have 2 safety visits and 4 assessment visits. Each Assessment visit will involve clinical tests, a blood test and an MRI scan. Healthy Volunteers will be recruited and undergo a screening visit and MRI scan.

ELIGIBILITY:
Inclusion criteria for AD:

* Subjects aged between 60-90 years old
* Male or postmenopausal female
* Fertile men are eligible to participate if they are willing to use the contraception methods listed in the PIS, during treatment and for 90 days after the last dose of treatment
* Able to provide written informed consent prior to any study-mandated procedures
* AA genotype at rs6971 (TSPO) locus
* Clinical diagnosis of AD by dementia specialist, fulfilling NIA-AA criteria
* Mild - moderate cognitive impairment (MMSE = 20-27 )
* AD biomarker positive MCI patients

Inclusion criteria for HV:

* Subjects aged 18 years or older
* Male or Female
* Female subjects of childbearing potential must be willing to have a pregnancy test before scanning
* Able to provide written informed consent prior to any study-mandated procedures
* Subjects willing to have blood samples collected for genotyping (ApoE and TSPO rs6971)
* AD biomarker positive

Exclusion criteria for AD:

* History of migraine (with attack frequency greater than 1 per month)
* Clinical history of suggestive of dementia with Lewy Bodies such as REM Sleep Behaviour Disorder
* Conditions affecting safe engagement in the intervention
* Conditions preventing completion of study procedures, e.g. severe loss of vision or hearing
* Clinically significant renal disease (eGFR <60 ml/min per 1.73m2)
* Clinically significant liver disease (abnormal serum transaminases)
* Contraindications to MRI scanning or exposure to gadolinium-based contrast agents
* Change of medications approved for AD (eg. Galantamine, rivastigmine, and donepezil) or antihypertensives within the last 28 days or planned during the timeframe of the study
* Severe respiratory disease with chronic hypoxia (sats <92%), known CO2 retention or need for home oxygen therapy
* Use of the following medications or therapies:
* Severe and moderate P450 CY3A4 inhibitors: Boceprevir, Clarithromycin, Cobicistat, Idelalisib, Itraconazole, Ketoconazole, Nelfinavir, Ritonavir, Saquinavir, Telaprevir, Telithromycin, Voriconazoleb, Aprepitant, Conivaptan, Crizotinib, Diltiazem, Dronedarone, Erythromycin, Fluconazole, Imatinib, Isavuconazole, Nefazodone, Netupitant, Nilotinib, Posaconazolee, Tofisopam, Verapamil, Delavirdine
* Severe and moderate P450 CY3A4 inducers: Carbamazepine, Enzalutamide, Fosphenytoin, Mitotane, Phenytoin, Rifampicin, Bosentan, Efavirenz, St John's wort, Barbiturates, Nevirapine, Primidone, Rifabutin, Rifapentine
* Oral contraceptives

Exclusion criteria for HV

* Contraindications to MRI scanning or exposure to gadolinium-based contrast agents
* Pregnancy in WOCBP
* eGFR<60 ml/min per 1.73 m2
* Severe respiratory disease with chronic hypoxia (sats <92%), known CO2 retention or need for home oxygen therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Does pharmacological modulation of TSPO (with XBD173, 90mg twice daily, orally, for 28 days) improve neurovascular coupling (NVC) in people with AD compared to placebo? | From baseline to 4 week follow-up after taking medication/placebo
  Does pharmacological modulation of TSPO (with XBD173, 90mg twice daily, orally, for 28 days) improve neurovascular coupling (NVC) in people with AD compared to placebo? NVC will be defined as the change in hippocampal cerebral blood flow (CBF) that follows a memory task (ΔCBF(h)).

CONTACTS AND LOCATIONS:
Overall Officials: David Owen, Principal Investigator — Imperial College London
Locations (1):
- NIHR Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No